CLINICAL TRIAL: NCT04985292
Title: Does Probiotic Supplementation Prevent Kidney Injury During Strenuous Physical Exercise?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2021-01332
Record Dates: First submitted 2021-06-10; First posted 2021-08-02 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Heat Stress; Kidney Injury
Keywords: Heat stress; Probiotic; Kidney Injury; Gut permeability
MeSH Terms: conditions — Heat Stress Disorders | interventions — Probiotics; Lacteol

STUDY DESIGN:
Intervention Model Description: Before each run (each study participant may only be included in one run) approximately half runners are randomized to receive a probiotic supplement and the other half to receive placebo
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The investigator will be provided with numbered boxes containing study products with identical probiotic and placebo capsules. The numbers have been generated using a block randomization (investigator blinded to length of block). Participants in each of the race will be allocated to receive one of the study product boxes depending on 1. Race order (all participants in the first race receive study product before any participant in the second race), and 2. Time of recruitment into study.
  There is no care provider in this study of healthy individuals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Probiotic (Experimental): 10^10 colony-forming units of a Lactobacillus strain, packaged in a capsule, once daily
  Interventions: Dietary Supplement: Probiotic, Lactobacillus
- Placebo (Placebo Comparator): Inactive substance packaged to be identical to active treatment
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic, Lactobacillus — 10^10 colony-forming units of a Lactobacillus strain, packaged in a capsule, once daily
  Arms: Probiotic
Dietary Supplement: Placebo — Inactive substance packaged to be identical to active treatment
  Arms: Placebo

SUMMARY:
Severe heat strain arising from intense physical work under climate conditions that does not allow sufficient heat dissipation may lead to heat stroke. This severe conditions is hypothesized to be secondary to increased gut permeability and leakage of bacterial toxins across the gut membrane, stimulating a systematic inflammatory response and associated organ injury. Repeated such sub-clinical increases in gut permeability has been suggested to contribute to the high burden of chronic kidney disease among heat-stressed workers. Many marathon runners experience a transient increase in kidney injury biomarkers while running. Probiotics have been studied as a way to decrease gut permeability and reduce systemic inflammation in many settings, including in athletes . However, no study has measured renal outcomes among workers or athletes performing strenuous activity. This is of interest as it could test the hypothesis that gut-induced inflammation is a driver of kidney injury during heat stress, and could point to a possible intervention to add on to efforts to relieve heat strain.

In the present study, recreational or professional runners will be randomized to take a probiotic supplement or placebo during a 4 week period preceding a strenuous physical exercise (minimum 21 km run). Urine samples will be taken before and after the run, and analyzed for markers of renal injury and inflammation.

DETAILED DESCRIPTION:
Participants registered to run in organised half-marathons, marathons and ultramarathons in Southern Sweden will be recruited. They will be asked to abstain from probiotic supplementation (including functional foods with probiotics) for 2 weeks, and then commence a 4-week period of probiotic or placebo supplementation.

At the end of the 4 week treatment period, the participants run the race. Urine samples are taken before and after the race and analysed for kidney injury markers.

Stool samples are taken by participants at the initiation of the treatment period, last stool before the race, and first stool after the race.

ELIGIBILITY:
Inclusion Criteria:

* Planning to run one of the long-distance races included.

Exclusion Criteria:

* Not having run at least 21 km previously,
* smoking,
* living too far away from the study area,
* unwilling to abstain from probiotic supplementation during treatment period,
* unwilling to abstain from NSAIDs or gut-permeability lowering supplements before the run,
* regular use of prescribed drugs (including hormonal contraceptives).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Urine tubular kidney injury marker (Kidney Injury Molecule 1 (KIM-1), monocyte chemotactic protein 1 (MCP-1), Insulin Growth Factor Binding Protein 7 (IGFBP-7)) composite variable aggregated using structural equations modelling. | From before the run to after the run (estimated run times 2-24 hours), morning urine after run, and 24 hours after the run finish. These time point are combined to one main outcome by calculating the area under the curve.
  Tubular injury markers measured in urine (e.g. KIM-1, MCP-1, IGFBP-7) combined using structural equations modelling and then combined over the 24 hour post-run period by calculating the area under the curve of this composite outcome variable in the 24 hours after the run. Exact list of markers to be determined based on budget available after sample collection is completed.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Jakobsson, MD, PhD, Principal Investigator — Göteborg University
Locations (1):
- Occupational and Environmental Medicine, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
No information that could be used to identify individuals will be shared. Considering the small size of the study and that it will most likely be conducted over multiple small runs, it is unlikely that any information on age and sex of participants could be shared without a risk of revealing the identity of the individual. Data on treatment allocation, biological measurement and questionnaire data without such identifying individual participant information will however be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the researchers have reported on the pre-specified research questions or otherwise have decided to make the data publicly available before this. This may be in approximately 2023-2024. We will keep the records for five years.
Access Criteria: Scientifically sound proposal.

REFERENCES:
- [Background] Mansour SG, Verma G, Pata RW, Martin TG, Perazella MA, Parikh CR. Kidney Injury and Repair Biomarkers in Marathon Runners. Am J Kidney Dis. 2017 Aug;70(2):252-261. doi: 10.1053/j.ajkd.2017.01.045. Epub 2017 Mar 28. PMID 28363731
- [Background] Hansson E, Glaser J, Jakobsson K, Weiss I, Wesseling C, Lucas RAI, Wei JLK, Ekstrom U, Wijkstrom J, Bodin T, Johnson RJ, Wegman DH. Pathophysiological Mechanisms by which Heat Stress Potentially Induces Kidney Inflammation and Chronic Kidney Disease in Sugarcane Workers. Nutrients. 2020 Jun 2;12(6):1639. doi: 10.3390/nu12061639. PMID 32498242
- [Background] Leon LR, Bouchama A. Heat stroke. Compr Physiol. 2015 Apr;5(2):611-47. doi: 10.1002/cphy.c140017. PMID 25880507
- [Background] Vaisberg M, Paixao V, Almeida EB, Santos JMB, Foster R, Rossi M, Pithon-Curi TC, Gorjao R, Momesso CM, Andrade MS, Araujo JR, Garcia MC, Cohen M, Perez EC, Santos-Dias A, Vieira RP, Bachi ALL. Daily Intake of Fermented Milk Containing Lactobacillus casei Shirota (Lcs) Modulates Systemic and Upper Airways Immune/Inflammatory Responses in Marathon Runners. Nutrients. 2019 Jul 22;11(7):1678. doi: 10.3390/nu11071678. PMID 31336570